CLINICAL TRIAL: NCT00694889
Title: Randomized Clinical Trial of Intensive Computer-based Cognitive Remediation in Recent-onset Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06TAF-972
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
Keywords: Psychosis; First Episode; Schizophrenia; Cognitive Remediation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Participants will use commercially available computer games.
  Interventions: Behavioral: Computer games
- 2 (Experimental): Participants will receive targeted cognitive training with neuroplasticity-based software created by Posit Science Corporation.
  Interventions: Behavioral: Neuroadaptive cognitive training
- 3 (Active Comparator): Healthy participants will receive targeted cognitive training with neuroplasticity-based software created by Posit Science Corporation.
  Interventions: Behavioral: Neuroadaptive cognitive training

INTERVENTIONS:
Behavioral: Neuroadaptive cognitive training — Neuroadaptive cognitive training includes cognitive remediation exercises that participants will practice 1 hour per day, 5 days per week, for 8 weeks. The exercises are specifically designed to improve speed and accuracy in the perception of and response to verbal targets. The treatment will focus on TCT.
  Arms: 2; 3
Behavioral: Computer games — The control treatment involves commercially available computer games that participants will practice 1 hour per day, 5 days per week, for 16 weeks.
  Arms: 1

SUMMARY:
The aim of this study is to investigate the efficacy of neuroscience-guided computerized cognitive training exercises on the remediation of cognitive deficits and symptoms associated with recent-onset schizophrenia and to examine the influence of subject characteristics, brain structure and function, and pharmacotherapy on the response to remediation.

DETAILED DESCRIPTION:
Participation in this study will last approximately 12 months and will involve individuals with recent-onset schizophrenia. All participants will undergo baseline assessments that will include an interview, written tests, blood draws, and electroencephalogram (EEG) and magnetic resonance imaging (MRI) scans. Participants will then be assigned randomly to receive treatment with either computerized neuroadaptive cognitive training or commercially available computer games. Participants will be asked to complete 60-minute sessions of their assigned treatments 5 days per week for 8 weeks. For participants receiving cognitive training, exercises will focus on improving speed and accuracy in the perception of and response to verbal and visuospatial targets. The 8 weeks of treatment will focus on targeted cognitive training (TCT). Participants assigned to practice computer games will play standard commercially available games, with no targeted response.

Participants will repeat baseline assessments after the computer training and Month 6 of follow-up. The EEG and MRI will be repeated only at post training assessment visit. There will be a blood draw at Week 2 of treatment as well. After the Month 6 assessment, participants in the control condition will be offered an opportunity to complete an additional 8 weeks of computer training with different modules.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder
* First psychotic episode within the last 3 years
* Good general physical health
* Age between 12-35
* Is fluent and proficient in the English language
* Achieved clinical stability (e.g., outpatient status for at least 3 months before study entry; on stable doses of medication for at least 1 month before study entry
* Minors must have parental/legal guardian consent to participate

Exclusion Criteria:

* Any neurological disorder
* History of psychoactive substance abuse in the past 6 months

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2007-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance, as measured by a neuropsychological battery | Measured at Baseline, Week 8, and 6 Month Follow-Up

SECONDARY OUTCOMES:
Symptom profile, as measured by clinical interviews | Measured at Baseline, Week 8, and 6 Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of California, San Francisco; San Francisco VA Medical Center; NCIRE - The Veterans Health Research Institute; Rachel Loewy, PhD, Study Director — University of California, San Francisco; Cameron Carter, MD, Study Director — University of California, Davis
Locations (2):
- United States (2):
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Derived] Puig O, Fisher M, Loewy R, Miley K, Ramsay IS, Carter CS, Ragland JD, Niendam T, Vinogradov S. Early- Versus Adult-Onset Schizophrenia as a Predictor of Response to Neuroscience-Informed Cognitive Training. J Clin Psychiatry. 2020 Mar 3;81(2):18m12369. doi: 10.4088/JCP.18m12369. PMID 32141724
- [Derived] Roach BJ, Ford JM, Biagianti B, Hamilton HK, Ramsay IS, Fisher M, Loewy R, Vinogradov S, Mathalon DH. Efference copy/corollary discharge function and targeted cognitive training in patients with schizophrenia. Int J Psychophysiol. 2019 Nov;145:91-98. doi: 10.1016/j.ijpsycho.2018.12.015. Epub 2018 Dec 29. PMID 30599145
- [Derived] Biagianti B, Roach BJ, Fisher M, Loewy R, Ford JM, Vinogradov S, Mathalon DH. Trait aspects of auditory mismatch negativity predict response to auditory training in individuals with early illness schizophrenia. Neuropsychiatr Electrophysiol. 2017;3:2. doi: 10.1186/s40810-017-0024-9. Epub 2017 Jun 9. PMID 28845238
- [Derived] Biagianti B, Fisher M, Neilands TB, Loewy R, Vinogradov S. Engagement with the auditory processing system during targeted auditory cognitive training mediates changes in cognitive outcomes in individuals with schizophrenia. Neuropsychology. 2016 Nov;30(8):998-1008. doi: 10.1037/neu0000311. Epub 2016 Sep 12. PMID 27617637
- [Derived] Panizzutti R, Hamilton SP, Vinogradov S. Genetic correlate of cognitive training response in schizophrenia. Neuropharmacology. 2013 Jan;64(1):264-7. doi: 10.1016/j.neuropharm.2012.07.048. Epub 2012 Aug 7. PMID 22992330